CLINICAL TRIAL: NCT06740526
Title: A Phase 2b, Multicenter, Open-label, Single-arm Trial to Evaluate the Impact of Sibeprenlimab on Kidney Histopathology Through Repeat Kidney Biopsies in Adolescents and Adults With Immunoglobulin A Nephropathy
Brief Title: Trial of the Impact of Sibeprenlimab on Immunoglobulin A Nephropathy Kidney Tissue
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 417-201-00060
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-12

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sibeprenlimab (Experimental)
  Interventions: Drug: Sibeprenlimab

INTERVENTIONS:
Drug: Sibeprenlimab — Sibeprelimab SC (Period 1)
  Sibeprelimab SC (Period 2)

SUMMARY:
This is a phase 2b open-label trial to characterize histopathological biomarkers of disease in immunoglobulin A nephropathy (IgAN) and demonstrate potential changes in response to sibeprenlimab.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 16 years of age or older at the time of signing the informed consent/assent.
2. Source-verified kidney biopsy confirmed diagnosis of IgAN.
3. Participant has estimated glomerular filtration rate (eGFR) > 45 mL/min/1.73 m2 using serum creatinine (Chronic Kidney Disease-Epidemiology Collaboration [CKD EPI] creatinine eGFR 2021 equation for those 18 years and older; Chronic Kidney Disease in Children under age 25 [CKiD U25] eGFR equation for those younger than 18 years)

Exclusion Criteria:

1. Participants who are breast-feeding and/or who have a positive pregnancy test result prior to receiving sibeprenlimab.
2. Participant has coexisting chronic kidney disease, other than IgAN.
3. Participant has a serum IgG value <600 mg/dL at screening.
4. Participant is currently receiving or has received within 24 weeks prior to the firstdose of sibeprenlimab, systemic corticosteroids or immunosuppression (note:

   topical, ophthalmic, rectal, intra-articular, inhaled corticosteroids are allowed).
5. Participant has uncontrolled hypertension (defined as systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg).
6. Participants who would be likely to require prohibited concomitant therapy during the trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2029-04-17 (Estimated); Study Completion 2029-04-17 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Glomerular IgA Deposition by Immunofluorescence in Kidney Tissue to Week 52 | From Baseline to Week 52

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Clinical Research Site 330, Denver, Colorado
  - Clinical Research Site 369, Boston, Massachusetts
  - Clinical Research Site 374, Dakota Dunes, South Dakota
  - Clinical Research Site 324, Houston, Texas
- Clinical Research Site 305, Scarborough Village, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: http://clinical-trials.otsuka.com